CLINICAL TRIAL: NCT03283306
Title: Prognostic Value of Carotid Contrast-Enhanced Ultrasound in Acute Ischemic Stroke Patients for Cerebrovascular and Cardiovascular Event
Brief Title: Prognostic Value of Carotid CEUS in Acute Ischemic Stroke Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other); Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Yeo Koon Kim, Assistant Professor, Seoul National University Hospital
Other Study IDs: B-1607-356-304
Record Dates: First submitted 2017-09-11; First posted 2017-09-14 (Actual); Last update posted 2017-09-14 (Actual); Status verified 2017-09

CONDITIONS: Ultrasonography; Carotid Stenosis; Ischemic Stroke
MeSH Terms: conditions — Carotid Stenosis; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Contrast-enhanced ultrasound(CEUS) of carotid artery plaque is a novel method that enabled direct visualization of neovessels in the vulnerable plaque. Plaque enhancement with CEUS showed correlation with the histologic density of neovessels within the carotid plaque and the previous cardiovascular events. Vulnerable plaques with a high risk of thromboembolic complications and rapid progression is associated with acute ischemic stroke. The prognostic value of vulnerable carotid artery plaque depicted with CEUS has not been fully investigated. The purpose of this study is to define prognostic value of plaque enhancement on carotid CEUS in acute stroke patients. Research question is; in acute ischemic stroke patients with ipsilateral carotid plaque as probable etiology of stroke, is the presence of carotid plaque enhancement on CEUS independent predictor of future stroke.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 19 years presenting acute ischemic stroke.
2. Compatible neurologic symptom within 14 days
3. Compatible MRI finding (one or more positive DWI lesions in the territory of unilateral ICA: ACA or MCA territory) - interpretable MRI image obtained in SNUBH or outside hospital
4. Etiology of acute ischemic stroke: except cardioembolic stroke (Atrial fibrillation) and other determined etiology
5. Ipsilateral extracranial carotid artery stenosis on MRA (CE-MRA), CTA or Doppler ultrasound

Exclusion Criteria:

1. History of ipsilateral carotid stent or endarterectomy
2. Carotid intervention during hospital stay
3. Contraindication to ultrasound contrast agent (SonoVue) A. Right to left, bi-directional, or transient right to left cardiac shunts B. History of hypersensitivity reactions to sulfur hexafluoride lipid microsphere components or any ultrasound contrast agent C. Pregnant or lactating woman D. Unstable cardiopulmonary conditions (acute myocardial infarction, acute coronary artery syndromes, worsening congestive heart failure, or serious ventricular arrhythmias)
4. Expected life span less than 12 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized acute ischemic stroke patients with ipsilateral carotid artery stenosis.
Sampling Method: Non-Probability Sample
Enrollment: 667 (Estimated)
Dates: Start 2017-08-09 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Composite of recurrent stroke, vascular death and myocardial infarction | 12 months
  (1) recurrent stroke: newly appeared DWI positive lesion on brain MRI with corresponding neurologic symptom (2) vascular death: sudden death, death due to stroke, myocardial infarction, heart failure, arrhythmia, pulmonary embolism, systemic bleeding, or ischemia of organ. (3) myocardial infarction: at least two of the followings: ① a history of typical angina pain. ② Elevation of Troponin, ③ Newly developed ST change or Q waves or LBBB on ECG (outcomes will be measured by chart review or physician diagnosis or telephone interview)

SECONDARY OUTCOMES:
Ipsilateral stroke | 12 months
  Recurrent stroke of ipsilateral side (recurrent stroke at same side of previous infarction)
All-cause mortality | 12 months
  All of the deaths, regardless of the cause
Carotid intervention | 12 months
  Ipsilateral carotid endarterectomy or carotid artery stent insertion which was not planned when discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Yeo Koon Kim, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided